CLINICAL TRIAL: NCT04067011
Title: A Phase 2 Drug-Vaccine Interaction Study to Examine Whether Co-administering AV7909 With Ciprofloxacin or Doxycycline Affects Antibiotic Pharmacokinetics or AV7909 Immunogenicity in Healthy Adults
Brief Title: Velocity 2: An Anthrax Vaccine and Antibiotics Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBS.AVA.210
Record Dates: First submitted 2019-07-15; First posted 2019-08-26 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Anthrax
Keywords: Antibiotics; Pharmacokinetics; Vaccine; Ciprofloxacin; Doxycycline; CPG 7909; Bacillus anthracis; Anthrax Vaccine Adsorbed; Post-exposure Prophylaxis; Adjuvant
MeSH Terms: conditions — Anthrax | interventions — Ciprofloxacin; Tablets; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1:Ciprofloxacin + AV7909 (Experimental): Participants meeting entry criteria will be randomized 1:1:1 to one of three investigational study groups. Groups 1 to 3 will each receive a manufactured lot of AV7909 per the study visit schedule.
  Group 1 will concomitantly receive ciprofloxacin.
  Interventions: Drug: Ciprofloxacin 500Mg Tablet; Biological: AV7909
- Group 2: Doxycycline +AV7909 (Experimental): Participants meeting entry criteria will be randomized 1:1:1 to one of three investigational study groups. Groups 1 to 3 will each receive a manufactured lot of AV7909 per the study visit schedule.
  Group 2 will concomitantly receive doxycycline.
  Interventions: Drug: Doxycycline 100Mg Tablet; Biological: AV7909
- Group 3: AV7909 (Experimental): Participants meeting entry criteria will be randomized 1:1:1 to one of three investigational study groups. Groups 1 to 3 will each receive a manufactured lot of AV7909 per the study visit schedule.
  Interventions: Biological: AV7909

INTERVENTIONS:
Drug: Ciprofloxacin 500Mg Tablet — Ciprofloxacin 500mg administered by mouth every 12 hours. The antibiotic will be administered orally on Study Days 4-9, 22-24 and 31-37.
  Arms: Group 1:Ciprofloxacin + AV7909
Drug: Doxycycline 100Mg Tablet — Doxycycline 100mg administered by mouth every 12 hours. The antibiotic will be administered orally on Study Days 2-9, 22-24 and 32-38.
  Arms: Group 2: Doxycycline +AV7909
Biological: AV7909 — 0.5mL AVA and 0.25mg CPG 7909 per 0.5mL dose.The vaccine will be administered intramuscularly on Study Days 8 and 23.

SUMMARY:
This study is designed to evaluate the pharmacokinetic (PK) profiles of ciprofloxacin or doxycycline when administered orally, prior to, and following, the intramuscular (IM) administration of a two-dose schedule of AV7909 administered two weeks apart.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multicenter, randomized trial designed to evaluate the pharmacokinetic profile, immunogenicity, and safety of AV7909 and ciprofloxacin or doxycycline when administered concomitantly in healthy adults for an indication of post-exposure prophylaxis (PEP) of anthrax.

Healthy adults between 18 to 45 years of age (inclusive) will sign and date an informed consent form and then be screened for eligibility for participation in the study 2 to 28 days prior to randomization. Participants meeting the entry criteria will be randomized 1:1:1 to one of the three study groups (AV7909 + ciprofloxacin, AV7909 + doxycycline and AV7909 only) on Day 1.

Subjects randomized into Groups 1 & 2 will be assigned to subgroups. Subgroup A will be assigned to the antibiotic PK treatment group first, while subgroup B will be assigned to the antibiotic non-PK treatment group.

Participants will be evaluated for safety through Day 51 [or the early withdrawal visit (EWV)], as assessed by clinical laboratory tests (hematology, serum chemistry, and urinalysis), monitoring of Adverse Events (AEs) including Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs), vital signs, and physical examinations. Adverse Events of Special Interest are adverse events associated with autoimmune disease as defined by the Center for Biologics Evaluation and Research, and might represent a safety signal for vaccine-associated autoimmunity. Reactogenicity (solicited systemic and injection site reactions) will be assessed daily by the participants using electronic diaries (e-diaries) after each vaccination. The e-diary will also be used to record self-administration of antibiotics for applicable study groups.

Information on the use of medications will be collected at each study visit. In addition, blood samples for auto-antibody assessment will be taken at Day 1 pre-dose and Day 51 (or Early Withdrawal Visit).

Participants who receive at least one dose of vaccine will also be asked to participate in safety follow-up phone calls occurring on Month 3, Month 6, Month 9, and Month 12 (nominally 3, 6, 9, and 12 months after the last vaccination) to collect information on AEs, SAEs and any potential AESIs. Based on responses at these phone contacts, participants may be asked to return to the clinic for an unscheduled visit to provide blood samples for auto-antibody testing to investigate reports of potential AESIs.

Independent safety oversight will be provided by a Data Safety Monitoring Board, which will be notified of significant AEs, potential AEsIs, or any other events as determined by the Medical Monitor, on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the participant (dated, signed, and captured in the medical chart at the site).
2. A male or female, aged 18 to 45 years of age, inclusive, at the time of informed consent.
3. Healthy condition as established by medical history and clinical examination before entering into the study.
4. Body mass index (BMI) less than or equal to 35.0 kg/m^2 at the Screening visit.
5. Have adequate venous access for phlebotomies.
6. For a woman of childbearing potential (WOCBP), negative pregnancy test at Screening and pre-randomization on Day 1, not currently breastfeeding, and no intention to become pregnant during the study period through 12 months after last receipt of any investigational product (IP). Every female participant is considered to be a WOCBP unless she is surgically sterile (hysterectomy, bilateral salpingectomy or bilateral oophorectomy) OR postmenopausal (defined as >12 consecutive months without menses and screen follicle-stimulating hormone > 30 mIU/mL). Women who are not of childbearing potential are allowed to enroll if they are surgically sterile or postmenopausal as defined above.

Female participants randomized to Groups 1 or 2 must be willing to add a double-barrier method, IUD, or abstinence as back-up forms of birth control since ciprofloxacin and doxycycline may decrease the effectiveness of birth control pills, implantable or injectable contraceptives.

Exclusion Criteria:

1. A Screening clinical laboratory test result greater than the central laboratory's upper limit of normal (ULN) for aspartate aminotransferase (AST), alanine aminotransferase (ALT), random glucose, total bilirubin, blood urea nitrogen (BUN), or creatinine. Other serum chemistry parameters that are not within the reference range will not be considered exclusionary unless deemed clinically significant by the principal investigator.
2. History of allergic reaction or intolerance to quinolone antimicrobials or any medical condition that would contraindicate the use of ciprofloxacin, including and not limited to vascular disorders, tendon disorders, certain genetic connective tissue disorders (e.g., Marfan and Ehlers-Danlos syndrome), prolongation of QT interval, seizures, peripheral neuropathy, increased risk of C. difficile infection.
3. History of allergic reaction or intolerance to tetracycline antibiotics or any medical condition that would contraindicate the use of doxycycline including an increased risk of C. difficile infection, increases in BUN or an increased sensitivity to direct sunlight or ultraviolet radiation resulting in erythema.
4. Has a need for any of the prohibited medications or requires the medications/foods within the prohibited times.
5. Have a tattoo/scar/birthmark or any other skin condition affecting the deltoid area that may interfere with injection site assessments.
6. History of anthrax disease, suspected exposure to anthrax, or previous vaccination with any anthrax vaccine.
7. Have previously served in the military any time after 1990 or plan to enlist in the military any time from Screening through the final telephone contact.
8. Previous anaphylactic reaction, severe systemic response, or serious hypersensitivity to a prior immunization or a known allergy to synthetic ODNs, aluminum, formaldehyde, benzethonium chloride (phemerol).
9. Plan to have an elective surgery at any point during the study until after the final safety phone contact.
10. Have donated or plan to donate blood within one month prior to enrollment or at any point during the study until after the final safety phone contact.
11. Use of any investigational or non-registered product (drug, vaccine or biologic) within 30 days preceding the dose of study vaccine, or planned use during the study until after the final safety phone contact.
12. Planned administration of any commercially-available vaccine from one week prior to the first study vaccination through two weeks after the last vaccination.
13. Have experienced chronic dosing (defined as more than 14 days) with any immune-modifying drugs within six months of study enrollment. This includes oral, intramuscular, intra-articular, intravenous, or inhalation corticosteroids except in the case of inhaled or intranasal medications for seasonal allergies.
14. Receipt of immunoglobulins and/or any blood products within the three months preceding study enrollment or at any point during the study period until after the final safety visit on Day 51.
15. An abnormal electrocardiogram (ECG) at screening interpreted as 'Abnormal, Significant'. Inclusion of participants with 'Abnormal, Insignificant' ECGs will be based on the principal investigator's discretion.
16. Have an active malignancy or history of metastatic or hematologic malignancy.
17. Have a history of an autoimmune, inflammatory, vasculitic or rheumaticor rheumatic disease including but not limited to systemic lupus erythematosus, Guillain-Barré syndrome, myasthenia gravis, polymyalgia rheumatica, diabetes mellitus type I, rheumatoid arthritis or scleroderma.
18. A positive laboratory evidence of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) HIV-1 or HIV-2 infection.
19. Positive result on urine drug screen, any evidence of ongoing drug abuse or dependence (including alcohol), or recent history (over the past five years) of treatment for alcohol or drug abuse.
20. Has an acute disease at the time of enrollment.
21. Any medical condition that, in the opinion of the investigator, could adversely impact the participant's involvement or the conduct of the study.
22. Have a significant chronic condition, e.g., serious cardiovascular, pulmonary, hepatic, type II diabetes mellitus or renal disease that, in the opinion of the investigator, would render treatment unsafe or would interfere with trial evaluations or completion of the study.
23. An opinion of the investigator that it would be unwise to allow the participant to be randomized into the study.
24. Member or immediate family member of an investigator site team.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Drobic, Study Director — Emergent BioSolutions
Locations (4):
- United States (4):
  - Avail Clinical Research, LLC, DeLand, Florida
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - New Orleans Center for Clinical Research / Volunteer Research Group, Knoxville, Tennessee

REFERENCES:
- [Derived] Drobic B, Akintunde G, Kim J, Mirceta M, Beach M, Komlenovic V. Effect of Co-administration of the anthrax vaccine adsorbed, adjuvanted with ciprofloxacin or doxycycline on antibiotic pharmacokinetics and the vaccine immunogenicity: A phase 2 drug-vaccine interaction study. Vaccine. 2026 Feb 15;73:128135. doi: 10.1016/j.vaccine.2025.128135. Epub 2025 Dec 24. PMID 41447782

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1:Ciprofloxacin + AV7909: Group 1 concomitantly received ciprofloxacin and AV7909.
  Ciprofloxacin 500Mg Tablet: Ciprofloxacin 500mg was administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 4-9, 22-24 and 31-37.
  AV7909: 0.5mL AVA and 0.25mg CPG 7909 per 0.5mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
- Group 2: Doxycycline +AV7909: Group 2 concomitantly received doxycycline and AV7909.
  Doxycycline 100mg Tablet: Doxycycline 100mg was administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 2-9, 22-24 and 32-38.
  AV7909: 0.5mL AVA and 0.25mg CPG 7909 per 0.5mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
- Group 3: AV7909: AV7909: 0.5mL AVA and 0.25mg CPG 7909 per 0.5mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
Period: Overall Study
Arm/Group | Group 1:Ciprofloxacin + AV7909 | Group 2: Doxycycline +AV7909 | Group 3: AV7909
Started | 70 | 71 | 69
Completed | 51 | 58 | 61
Not Completed | 19 | 13 | 8
Not completed — Not Treated | 8 | 7 | 5
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Other Reasons | 2 | 0 | 1
Not completed — Missing | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population: all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1:Ciprofloxacin + AV7909 | Group 2: Doxycycline +AV7909 | Group 3: AV7909 | Total
Number analyzed (Participants) | 70 | 71 | 69 | 210
Age, Customized [Count of Participants; unit: Participants]
  18 - 30 years | 29 | 30 | 31 | 90
  31 - 45 years | 41 | 41 | 38 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 47 | 43 | 134
  Male | 26 | 24 | 26 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 20 | 26 | 17 | 63
  White | 46 | 43 | 48 | 137
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 70 | 71 | 69 | 210
Height [Mean (Standard Deviation); unit: cm] | 170.1 (9.8) | 169.1 (8.5) | 169.7 (10.7) | 169.6 (9.7)
Weight [Mean (Standard Deviation); unit: kg] | 78.7 (16.7) | 79.4 (12.6) | 75.0 (16.0) | 77.7 (15.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.9) | 27.7 (3.7) | 25.9 (4.6) | 26.9 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Ciprofloxacin Area Under the Curve From 0 to 12 Hours (AUC0-12h) and Maximum Concentration (Cmax) on Days 8 and 35
Description: Based on serum concentrations of ciprofloxacin on Day 8 (pre-AV7909 vaccination) and on Day 35 (post-AV7909 vaccination), steady state AUC0-12h and Cmax were derived, and geometric mean of ratio of AUC0-12h on Day35/Day 8 and geometric mean of ratio for Cmax on Day 35/Day8, and the corresponding 90% CI of the mean ratios were calculated.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours post-ciprofloxacin dose on Days 8 (pre-AV7909 vaccination) and 35 (post-AV7909 vaccination)
Population: The number of analyzed participants represents the number of participants that met pre-specified protocol criteria for inclusion in the PK analysis population.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Ciprofloxacin + AV7909: Participants meeting entry criteria were randomized 1:1:1 to one of three investigational study groups. Groups 1 to 3 each received a manufactured lot of AV7909 per the study visit schedule.
  Group 1 concomitantly received ciprofloxacin.
  Ciprofloxacin 500Mg Tablet: Ciprofloxacin 500mg administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 4-9, 22-24 and 31-37.
Arm/Group | Ciprofloxacin + AV7909
Number analyzed (Participants) | 25
Ratio
  Ratios of AUC0-12h (Post-vac./Pre-vac) | 0.9764 [0.8895 to 1.0718]
  Ratios of Cmax (Post-vac./Pre-vac) | 0.9706 [0.8693 to 1.0838]
Statistical Analysis 1: Comparison: Ciprofloxacin + AV7909; Analysis of Geometric mean ratio of area under the curve from 0 to 12 hours (AUC0-12h) for ciprofloxacin on Days 8 and 35; Test type: Equivalence — The equivalence testing was constructed using paired two one-sided t-tests (TOST) with natural log transformation of PK parameters. Results obtained from transformed analyses were back-transformed by exponentiation for presentation of the point estimates and 90% CIs for geometric mean ratio of AUC0-12h; Ratio of AUC = 0.9764, 90% CI 2-sided [0.8895 to 1.0718]
Statistical Analysis 2: Comparison: Ciprofloxacin + AV7909; Analysis of Geometric mean ration of Cmax for ciprofloxacin on Days 8 and 35; Test type: Equivalence — The equivalence testing was constructed using paired two one-sided t-tests (TOST) with natural log transformation of PK parameters. Results obtained from transformed analyses were back-transformed by exponentiation for presentation of the point estimates and 90% CIs for geometric mean ratio of Cmax; Ratio of Cmax = 0.9706, 90% CI 2-sided [0.8693 to 1.0838]

2. Primary Outcome: Ratio of Doxycycline Area Under the Curve From 0 to 12 Hours (AUC0-12h) and Maximum Concentration (Cmax) on Days 8 and 38
Description: Based on serum concentrations of doxycycline on Day 8 (pre-AV7909 vaccination) and on Day 38 (post-AV7909 vaccination), steady state AUC0-12h and Cmax were derived, and geometric mean of ratio of AUC0-12h on Day38/Day 8 and geometric mean of ratio for Cmax on Day 38/Day8, and the corresponding 90% CI of the mean ratios were calculated.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10 and 12 hours post-doxycycline dose on Days 8 (pre-AV7909 vaccination) and 38 (post-AV7909 vaccination)
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- Doxycycline + AV7909: Group 2 concomitantly received doxycycline. Doxycycline 100mg Tablet: Doxycycline 100mg was administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 2-9, 22-24 and 32-38.
  AV7909: 0.5mL AVA and 0.25mg CPG 7909 per 0.5mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
Arm/Group | Doxycycline + AV7909
Number analyzed (Participants) | 31
Ratio
  Ratios of AUC0-12h (Post-vac./Pre-vac) | 0.9173 [0.8187 to 1.0278]
  Ratios of Cmax (Post-vac./Pre-vac) | 0.8974 [0.7841 to 1.0271]
Statistical Analysis 1: Comparison: Doxycycline + AV7909; Analysis of Geometric mean ratio of Area under the curve from 0 to 12 hours (AUC0-12h) for doxycycline on Days 8 and 38; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of AUC = 0.9173, 90% CI 2-sided [0.8187 to 1.0278]
Statistical Analysis 2: Comparison: Doxycycline + AV7909; Analysis of Geometric mean ration of Cmax for doxycycline on Days 8 and 38; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of Cmax = 0.8974, 90% CI 2-sided [0.7841 to 1.0271]

3. Secondary Outcome: Geometric Mean TNA 50% Neutralizing Factor (NF50) Values Two Weeks After the Second AV7909 Vaccination (Day 37 ± 1 Day).
Description: Immunogenicity response as assessed by geometric mean of TNA NF50 values at Day 37 (two weeks after second dose of AV7909 vaccination).
Time Frame: Day 37 ± 1 day
Population: The number of analyzed participants represents the number of participants that met pre-specified protocol criteria for inclusion in the immunogenicity analysis population.
Measure: Geometric Mean (95% Confidence Interval); unit: TNA NF50 titer
Groups:
- Group 1:Ciprofloxacin + AV7909: Group 1 concomitantly received ciprofloxacin. Ciprofloxacin 500Mg Tablet: Ciprofloxacin 500mg was administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 4-9, 22-24 and 31-37.
  AV7909: 0.5mL AVA and 0.25mg CPG 7909 per 0.5mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
- Group 2: Doxycycline +AV7909: Group 2 concomitantly received doxycycline. Doxycycline 100mg Tablet: Doxycycline 100mg was administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 2-9, 22-24 and 32-38.
  AV7909: 0.5mL AVA and 0.25mg CPG 7909 per 0.5mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
Arm/Group | Group 1:Ciprofloxacin + AV7909 | Group 2: Doxycycline +AV7909 | Group 3: AV7909
Number analyzed (Participants) | 47 | 50 | 54
TNA NF50 titer | 1.8 [1.3 to 2.4] | 1.8 [1.4 to 2.3] | 1.6 [1.3 to 2.0]
Statistical Analysis 1: Comparison: Group 1:Ciprofloxacin + AV7909 vs Group 3: AV7909; Test type: Non-Inferiority — Non-inferiority margin is 0.5; Ratio of GMT (Group 1/Group 3) = 1.13, 95% CI 2-sided [0.78 to 1.64]
Statistical Analysis 2: Comparison: Group 2: Doxycycline +AV7909 vs Group 3: AV7909; Test type: Non-Inferiority — Non-inferiority margin is 0.5; Ratio of GMT (Group 2/Group 3) = 1.14, 95% CI 2-sided [0.81 to 1.6]

ADVERSE EVENTS:
Time Frame: Incidence of adverse events (AEs) from the first dose of any study treatment (either antibiotic and/or AV7909 vaccine) through the Final Study Visit (Day 51 ± 1 day)
Description: Safety in all groups were assessed up to Day 51 (last in-clinic visit) by collecting adverse events (AEs; including serious adverse event), local and systemic reactogenicity events and assessments of physical examinations, vital signs, clinical laboratories (hematology, serum chemistry, urinalysis). Only participants that received at least one dose of study treatment are included in the safety population (i.e., 62 participants in Group 1; 64 participants in Group 2; 64 participants in Group 3).
Groups:
- Group 1: Ciprofloxacin + AV7909: Group 1 concomitantly received ciprofloxacin and AV7909.
  Ciprofloxacin 500 mg Tablet: Ciprofloxacin 500 mg administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 4-9, 22-24 and 31-37.
  AV7909: 0.5 mL AVA and 0.25mg CPG 7909 per 0.5 mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
- Group 2: Doxycycline +AV7909: Group 2 concomitantly received doxycycline and AV7909.
  Doxycycline 100 mg Tablet: Doxycycline 100 mg administered by mouth every 12 hours. The antibiotic was administered orally on Study Days 2-9, 22-24 and 32-38.
  AV7909: 0.5 mL AVA and 0.25mg CPG 7909 per 0.5 mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
- Group 3: AV7909: AV7909: 0.5 mL AVA and 0.25mg CPG 7909 per 0.5 mL dose. The vaccine was administered intramuscularly on Study Days 8 and 23.
Arm/Group | Group 1: Ciprofloxacin + AV7909 | Group 2: Doxycycline +AV7909 | Group 3: AV7909
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/62 | 0/64 | 1/64
Other Adverse Events (participants affected / at risk) | 17/62 | 17/64 | 16/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ciprofloxacin + AV7909 (N=62) | Group 2: Doxycycline +AV7909 (N=64) | Group 3: AV7909 (N=64)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ciprofloxacin + AV7909 (N=62) | Group 2: Doxycycline +AV7909 (N=64) | Group 3: AV7909 (N=64)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 2 (3)
Injection site pain (General disorders) | 6 (10) | 5 (11) | 8 (17)
Injection site induration (General disorders) | 2 (3) | 7 (8) | 5 (5)
Injection site movement impairment (General disorders) | 3 (3) | 2 (2) | 4 (5)
Vaccination complication (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 7 (9)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 4 (4) | 4 (6) | 4 (5)

LIMITATIONS AND CAVEATS:
No Limitations and Caveats in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT04067011/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04067011/SAP_001.pdf
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04067011/ICF_002.pdf